CLINICAL TRIAL: NCT06559800
Title: Step by Step - Pilot Study of Cognitive Behavior Therapy With Role-plays in Virtual Reality for Children With Anger, Oppositional or Aggressive Behaviors
Brief Title: Pilot Study of Cognitive Behavior Therapy With Role-plays in Virtual Reality for Children With Behavior Problems
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: PRIMA (Unknown); Psykologpartners (Unknown)
Responsible Party: Principal Investigator, Pia Enebrink, Associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00813-01 - Children
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Child Behavior Problem; Disruptive Behavior; Oppositional Defiant Disorder; Conduct Problems; Aggression; Anger
Keywords: Disruptive behavior; Child behavior problems; Cognitive behavior therapy; Virtual reality
MeSH Terms: conditions — Problem Behavior; Oppositional Defiant Disorder; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive behavior therapy for children and youth with role-plays in virtual reality (Experimental): Child/youth cognitive-behavioral program with up to 10 individual, face-to-face, weekly sessions
  Interventions: Behavioral: YourSkills: Cognitive behavioral therapy for children/youth with role-plays in virtual reality

INTERVENTIONS:
Behavioral: YourSkills: Cognitive behavioral therapy for children/youth with role-plays in virtual reality — A program for children/youth with anger problems or aggressive behaviors based on social learning theory and cognitive behavior therapy (CBT), incorporating virtual reality (VR) when conducting brief role-plays. The program includes similar strategies as other CBT-oriented programs for anger problems, with the addition of VR for practicing skills.

SUMMARY:
The main aim of this small pilot trial is to evaluate preliminary effects and feasibility of the child intervention YourSkills for child disruptive behavior (e.g., enhanced anger or aggressive behavior) when evaluated in Sweden for children/youth aged 10-16 years. YourSkills is based on cognitive behavioral therapy (CBT) and includes practicing of skills in virtual reality (VR).

The main questions the project aims to answer are:

* What are the preliminary effects of the child/youth CBT-VR-program?
* What is the level of child/youth engagement in the CBT-VR program?
* What are the experiences of parents, children/youth and therapists of the program?

The CBT-VR program is delivered at clinics during ten individual sessions. Parents will answer quantitative measurements before and after treatment, children will answer quantitative measurements before, during and after treatment. Within- group analyses will be conducted to examine experiences and preliminary effects of the program. Parents, children and clinicians are also asked to participate in a qualitative interview after the program has ended.

DETAILED DESCRIPTION:
Cognitive behavioral therapy (CBT) for children with behavior problems often include anger management training, social skills training, and problem-solving training. These have been shown to reduce anger and aggressive behaviors with small to moderate effects.

In a study in the Netherlands, the CBT-VR treatment program YourSkills was developed and evaluated for boys with aggressive behavior aged 8-13 years (Alsem et al, 2023). The treatment builds on CBT and includes brief role-plays conducted in virtual reality (VR). VR can provide a safe and gradual platform to practice.

PURPOSE AND RESEARCH QUESTIONS:

The aim of the pilot study is to evaluate preliminary effects and feasibility of the CBT-VR program YourSkills in Sweden for children/youth aged 10-16. The specific research questions are as follows:

1. What are the preliminary effects of the CBT-VR program on children's behavioral problems, well-being, parents' emotion regulation, parenting strategies, and family conflicts?
2. What is the level of child engagement in the CBT-VR program (e.g., the number of sessions, homework completion and dropout rates)?
3. What are the experiences of parents, children and therapists of the program (e.g., its effectiveness, acceptability, usefulness as well as relevance of the strategies taught)?

METHODS:

This project consists of a small pilot study of the CBT-based program YourSkills.

In the present project we target children/youth aged 10-16 years (n=10 families). The design is based on a mixed-methods approach. Evaluation of the intervention is conducted using within-group design (repeated measurements before, during, and after the intervention).

Families will be recruited through clinics and advertisements. They are directed to a webpage with information about the study and contact information to the researchers. Families provide informed consent to participate. Upon a participant expressing interest of the study, a member of the research team will contact the participant for a screening of inclusion and exclusion criteria.

The treatment is evaluated quantitatively by parents and children, using validated assessment scales before and after treatment, and by children with single questions before, during, and after the intervention. Additionally, qualitative interviews will be conducted with participants who consent to participate in an interview. Interviews will be recorded and transcribed. Clinicians at the clinics are invited to answer questions regarding their experiences of delivering the program.

In another separate pilot study we evaluate parent training with role-plays in virtual reality: "Pilot study of parent training with role-plays in virtual reality for parents of children with behavior problems".

POWER CALCULATION:

The quantitative and qualitative data that will be collected for ten families is considered sufficient to provide understanding and preliminary insight into acceptability, usability, relevance, and effectiveness.

ANALYSES:

The plan is to compare changes during the intervention using paired t-tests, descriptive statistics, description of reliable and clinical change, and calculation of effect sizes. If appropriate, non-parametric alternatives will be employed. The qualitative analyses will be conducted using content analysis or thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Child/youth aged between 10-16 years with increased levels of anger or disruptive behaviors,
* The child's behavior problems is elevated on questions targeting behavioral problems (SDQ conduct problems subscale).

Exclusion Criteria:

* Child/youth is below 10 years or above 16 years of age
* No increased levels of anger or disruptive behaviors
* Child/youth is diagnosed with autism, serious depression, psychosis, eating disorder, or self-harm behaviors
* Child/youth has epilepsy or migraine

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-08-19 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Parent: Mean change from baseline in behavior problems on parent-ratings of the Disruptive Behavior Disorder scale (oppositional defiant disorder subscale). | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  The oppositional defiant disorder subscale of the Disruptive Behavior Disorder scale is used for assessing children's behavioral problems. The subscale includes 8 items which are rated on a 4-point scale (0 to 3). The total scale sum ranges från 0 to a total maximum sum of 24 with a higher score indicating more behavior problems.
Child/youth: Mean change from baseline in child-ratings of anger on the Anger Expression Scale for children | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  The Anger expression scale for children includes 26 questions about anger and anger management and is rated by children on a 4-point Likert scale (from 1 to 4). We use two modified sub-scales: anger expression (score ranges from 17 to 68) and anger control (score ranges from 9 to 36) with higher scores indicating higher levels of anger expression and anger control.

SECONDARY OUTCOMES:
Parent: Mean change from baseline in parent-ratings of child wellbeing on the KIDSCREEN-10 | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  The KIDSCREEN has 10 items and evaluates how parents perceive the health and well-being of their child or adolescent. The items are scored on a 5-point scale (1-5). A total maximum sum ranges between 10 and 50, and a higher score indicates greater child wellbeing and health-related quality of life. The scale also includes an overall question about how the child is feeling in general.
Parent: Mean change from baseline in parent-ratings of child wellbeing on the Strengths and Difficulties Questionnaire (SDQ) | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  The Strengths and Difficulties Questionnaire (SDQ) assesses mental health through five subscales (peer relationship problems, prosocial behavior, emotional symptoms, hyperactivity/ inattention, conduct problems) and a total difficulties score. The items are scored on a 3-point scale (0 to 2), and the total difficulties score is generated by summing all subscales except the prosocial scale. The summary score ranges from 0 to 40 where higher summary scores indicate more problems.
Parent: Mean change from baseline in parent-ratings of emotion regulation on the Difficulties in Emotion Regulation Scale (brief version) | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  Parents' general emotion regulation ability will be measured with the Difficulties in Emotion Regulation Scale-16. The 16 items are scored on a 5-point scale (1 to 5). The total summary score ranges between 16 and 80, a higher score indicating larger difficulties with emotion regulation.
Parent: Mean change from baseline in parent-ratings of parental emotion regulation on the Parent Emotion Regulation Scale | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  Parental emotion regulation will be measured with Parent Emotion Regulation Scale. The 20 items are scored on a 5-point scale (1 to 5). A total summary score ranges between 20 and 100, with a higher score indicating better regulation of emotions.
Parent: Mean change in parent-ratings of family warmth | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  Family warmth is measured with 5 questions from the Family Check-Up Caregiver Assessment Scale. The items are scored on a 5-point scale (1 to 5). Total maximum score ranges between 5 and 25. A higher score indicates a more positive relation.
Parent: Mean change in parent-ratings of family conflicts | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  Three questions from the Family Check-Up Caregiver Assessment Scale are used to measure family conflicts. The items are scored on a 7-point scale (0 to 6), with total maximum score ranging between 0 and 18. A higher score indicates larger degree of conflicts.
Parent: Mean change from baseline in parenting on parent-ratings of the Parenting Children and Adolescents Scale | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  The three sub-scales of the Parenting Children and Adolescents Scale are Encouragement of positive behaviors; Setting limits; Proactive parenting behaviors. The 21 items are scored on a 5-point scale (1 to 5). The total scale sum ranges from 21 to a maximum of 105. A higher score indicates more positive parenting behaviors.
Parent: Mean change from baseline in parenting on parent-ratings of the Parenting Children and Adolescents Scale: Impact scale | Pre- and post-intervention (10 weeks after the initiation of the intervention)
  For each of the 21 items of the Parenting Children and Adolescents Scale the parent also indicates whether the item is experienced as a problem (yes/no). Total scale sum ranges between 0 and 21, with a higher sum indicating more problems and impact.
Child/youth: Mean change from baseline in child-ratings of child wellbeing on the Strengths and Difficulties Questionnaire | From pre- to post-intervention (measured after 10 weeks)
  Child-ratings of Strengths and Difficulties Questionnaire are used to assess mental health through a total difficulties score as well as through the five subscales (peer relationship problems, prosocial behavior, emotional symptoms, hyperactivity/inattention, conduct problems). The items are scored on a 3-point scale (0 to 2), and the total difficulties score is generated by summing all subscales except the prosocial scale. The summary score ranges from 0 to 40 where higher summary scores indicate more severe problems.
Child/youth: Mean change from baseline in child-ratings of child wellbeing on the KIDSCREEN-10 | From pre- to post-intervention (measured after 10 weeks)
  The instrument evaluates how children perceive their health and well-being. The 10 items are scored on a 5-point scale (1 to 5). The total maximum sum ranges between 10 and 50, with a higher score indicating greater child wellbeing and health- related quality of life. The scale also includes an overall question about how the child is feeling in general.
Child/youth: Satisfaction with the week | From pre- to post-intervention (during 10 weeks). Completed once a week at the session.
  One question rated 0-10 measuring satisfaction with the week. Higher levels indicate larger satisfaction.
Child/youth: Presence of anger or conflicts | From pre- to post-intervention (during 10 weeks). Completed once a week at the session.
  Two questions, each rated 0-10 (maximum score between 0- 20), measuring presence of anger or conflicts. Higher levels indicate larger anger problems/conflicts.
Child/youth: Child experiences of each session | From pre- to post-intervention (during 10 weeks). Completed once a week at the session
  Four questions after each session about how the child experienced the sessions and exercises. Rated on a scale 0-10, with a maximum total score ranging between 0 and 40. A higher score indicates greater satisfaction with the session.
Child/youth: Closing questions about the intervention | Post-intervention (10 weeks after the initiation of the intervention)
  Five closing questions about satisfaction, relevance, and usefulness of the intervention. The questions are rated on a 0-10-scale, total score is 50, with higher score indicating larger satisfaction.
Clinicians: Clinician perception of treatment implementation | From pre- to post-intervention (measured after 10 weeks)
  Clinicians conducting treatments will respond to two questions every week about treatment implementation. The questions are rated 0-10 (maximum weekly mean score 20), with higher scores indicating larger satisfaction.
Parent, child/youth, clinician: Experiences of the child/youth program through individual qualitative interviews with parent, youth or clinician | Interviews are conducted after the program is completed, about 10 weeks after the initiation of the program
  Qualitative interviews will explore parent's, child's/youth's and clinician's experiences of the treatment. We will investigate satisfaction, feasibility, acceptability, and relevance of the programs. The interview with parents is partly based on an established scale, modified for this purpose, and self-constructed questions. Interviews with clinicians and children are based on self-constructed questions examining acceptability, relevance, feasibility and satisfaction.
Use of the child/youth program: number of sessions, homework tasks | From pre- to post-intervention (10 weeks after the initiation of the intervention)
  A summary of the mean number of sessions and homework tasks completed during the program.
Drop-out rate | From pre- to post-intervention (10 weeks after the initiation of the intervention)
  The drop out from the program (number of participants)

OTHER OUTCOMES:
Background information - parent | Pre-intervention
  Parents are asked for brief demographic information about themselves (e.g., age, education) and their child (e.g. age). A total of 8 questions.
Background information - child | Pre-intervention
  Children are asked three demographic questions about themselves (e.g., age).

CONTACTS AND LOCATIONS:
Overall Officials: Pia Enebrink, PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alsem SC, van Dijk A, Verhulp EE, Dekkers TJ, De Castro BO. Treating children's aggressive behavior problems using cognitive behavior therapy with virtual reality: A multicenter randomized controlled trial. Child Dev. 2023 Nov-Dec;94(6):e344-e361. doi: 10.1111/cdev.13966. Epub 2023 Jul 17. PMID 37459452